CLINICAL TRIAL: NCT04983303
Title: Comparing The Effectiveness of Tracing Image and Coloring for Kids-Book With Two Active Distractions on Pain and Fear in Children During Venipuncture: A Randomized Controlled Trial
Brief Title: Comparison of the Effectiveness of Distraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Sherzad Khudeida Suleman, Principal Investigator, University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SRS
Record Dates: First submitted 2021-07-04; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Venipuncture
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TICK-B group as intervention group (Experimental): TICK-B group: The children will receive a picture as they want. They will be asked to trace and color the pictures that need coloring. After the procedure, the child will take his or her picture which he colored during the procedure.
  Interventions: Other: TICK-B group
- Coughing trick (Experimental): Coughing trick: Children in this group will be taught how to cough during the procedure. coughs with start moderate force and then coughs again which coincides with a needle procedure, such as venipuncture for example.
  Interventions: Other: TICK-B group
- Balloon inflation group as intervention group (Experimental): Balloon inflation group: In this group, the children will receive a balloon colored as their favorite, and they will be asked to inflate the balloon before starting the venipuncture procedure.
  Interventions: Other: TICK-B group
- Standard care provided group as control group (No Intervention): Standard care provided group as the control group

INTERVENTIONS:
Other: TICK-B group — These interventions will distract the child during venipuncture
  Other Names: Coughing trick group; Balloon inflation group; Control group or no intervention
  Arms: Balloon inflation group as intervention group; Coughing trick; TICK-B group as intervention group

SUMMARY:
Venipuncture, a frequently performed needle-related procedure, is one of the foremost frightening experiences, and a typical source of moderate to severe pain for pediatric patients.

No randomized studies have compared the effectiveness of balloon inﬂation, cough trick, and TICK-B on reducing pain in children between 6 and 12 years old during the drawing of venous blood samples. The research hypothesis was that children who draw and color a picture, inﬂate a balloon, or perform the cough trick while having their blood taken would experience less pain and anxiety than children who did not undergo a pain-reducing intervention.

Objectives:

To evaluate the roles of the TICK-B, balloon inflation, and cough trick in relieving pain and fear of school-age children during venipuncture.

To compare the effect of TICK-B with the effects of the cough trick, balloon inflation, on reducing pain and anxiety during venipuncture in children.

To compare the effects of three distraction groups with the control group in relieving pain and anxiety during venipuncture.

DETAILED DESCRIPTION:
Venipuncture, a frequently performed needle-related procedure, is one of the foremost frightening experiences, and a typical source of moderate to severe pain for pediatric patients. Approximately 83% of young children aged 2.5-6 years, 51% of youngsters aged 7-12 years, and 28% of adolescents (aged more than 12 years) who underwent venipuncture stated high levels of distress during the painful procedure. However, < 10% of venipuncture performing are given pain management.

To relieve pain, fear, and anxiety in children undergoing venipuncture or venous cannulation, both pharmacological and non-pharmacological approaches are used to help control pediatric patients' discomfort. Pain management includes pharmacologic and non-pharmacologic approaches. The most commonly used pharmacological approach to decrease medical procedure-related pain is the application of topical anesthetic creams. Non-pharmacological methods include distraction actions like blowing bubbles, reading, or playing a game.

Balloon inﬂation causes a reduction in venous return with increased intrathoracic pressure. It has been speculated that this increase in pressure induces baroreceptor activation with contraction of the pulmonary vessels and that the activation of cardiopulmonary and sinoaortic baroreceptor reﬂex arcs has an antinociceptive effect, resulting in pain relief.

Coughing increases intrathoracic pressure and stimulation to the autonomic nervous system, causing an increase in heart rate and blood pressure, a higher level of pressure in the subarachnoid space, and baroreceptor activation. The increase in pressure in the subarachnoid space activates the segmental pain inhibiting pathways; thus, the increase in blood pressure and baroreceptor activation appears to be efﬁcacious in reducing the perception of pain.

ELIGIBILITY:
Inclusion Criteria:

* School-aged 6-12 years old.
* Children who require venipuncture.

Exclusion Criteria:

1. Respiratory chronic diseases,
2. Physical impairment,
3. Disability contributing to difficult communication,
4. Children of unsatisfied parents,
5. Children with neurodevelopment delay,
6. Cognitive impairment, hearing impairment or a visual impairment,
7. Taking an analgesic within 6 hours, or for those with a syncope history.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Faces Pain Scale-Revised to rate the severity of Pain (0-10) from no pain to worst pain | 5 minutes before procedure done.
  To assess the intensity of pain related to the venipuncture procedure in children.
  Children will self-report their pain severity using the Faces Pain Scale-Revised, which has been validated and shown to be reliable.
Fear | 5 minutes before venipuncture procedure done
  To assess the fear level of the children related to the venipuncture procedure.
  Children will self-report their level of fear using the Children's Fear Scale (CFS), which has been validated and shown to be reliable.

SECONDARY OUTCOMES:
Faces Pain Scale-Revised to rate the severity of Pain (0-10) from no pain to worst pain | 0 minute during venipuncture procedure (time during insertion of cannula).
  To assess the intensity of pain related to venipuncture procedure in children:
  Children will self-report their pain severity using the Faces Pain Scale-Revised, which has been validated and shown to be reliable.
Faces Pain Scale-Revised to rate the severity of Pain (0-10) from no pain to worst pain. | 1-2 minute after venipuncture procedure done.
  To assess the intensity of pain related to the venipuncture procedure in children.
  Children will self-report their pain severity using the Faces Pain Scale-Revised, which has been validated and shown to be reliable.
Children's Fear Scale (CFS): Fear (0-4) no anxiety to extreme anxiety | 0 minute during venipuncture procedure.
  To assess the fear level of the children related to venipuncture procedure:
  -Children will self-report their level of fear using the Children's Fear Scale (CFS), which has been validated and shown to be reliable.
Children's Fear Scale (CFS): Fear (0-4) no anxiety to extreme anxiety | 1-2 minute after venipuncture procedure done.
  To assess the fear level of the children related to the venipuncture procedure:
  -Children will self-report their level of fear using the Children's Fear Scale (CFS), which has been validated and shown to be reliable.

OTHER OUTCOMES:
Visual Analog Scale (VAS), to measure the pain and Fear of children by the parents and observer. | Immediately after venipuncture (1-2 min.)
  Visual Analog Scale (VAS) will be used to measure pain and fear of children during venipuncture by parent and observer

REFERENCES:
- [Background] Stevens BJ, Abbott LK, Yamada J, Harrison D, Stinson J, Taddio A, Barwick M, Latimer M, Scott SD, Rashotte J, Campbell F, Finley GA; CIHR Team in Children's Pain. Epidemiology and management of painful procedures in children in Canadian hospitals. CMAJ. 2011 Apr 19;183(7):E403-10. doi: 10.1503/cmaj.101341. Epub 2011 Apr 4. PMID 21464171
- [Background] Walther-Larsen S, Pedersen MT, Friis SM, Aagaard GB, Romsing J, Jeppesen EM, Friedrichsdorf SJ. Pain prevalence in hospitalized children: a prospective cross-sectional survey in four Danish university hospitals. Acta Anaesthesiol Scand. 2017 Mar;61(3):328-337. doi: 10.1111/aas.12846. Epub 2016 Dec 29. PMID 28032329
- [Background] Taddio A, Appleton M, Bortolussi R, Chambers C, Dubey V, Halperin S, Hanrahan A, Ipp M, Lockett D, MacDonald N, Midmer D, Mousmanis P, Palda V, Pielak K, Riddell RP, Rieder M, Scott J, Shah V. Reducing the pain of childhood vaccination: an evidence-based clinical practice guideline (summary). CMAJ. 2010 Dec 14;182(18):1989-95. doi: 10.1503/cmaj.092048. Epub 2010 Nov 22. No abstract available. PMID 21098067
- [Background] Rogers TL, Ostrow CL. The use of EMLA cream to decrease venipuncture pain in children. J Pediatr Nurs. 2004 Feb;19(1):33-9. doi: 10.1016/j.pedn.2003.09.005. PMID 14963868
- [Background] Koller D, Goldman RD. Distraction techniques for children undergoing procedures: a critical review of pediatric research. J Pediatr Nurs. 2012 Dec;27(6):652-81. doi: 10.1016/j.pedn.2011.08.001. Epub 2011 Oct 13. PMID 21925588
- [Background] Gupta D, Agarwal A, Dhiraaj S, Tandon M, Kumar M, Singh RS, Singh PK, Singh U. An evaluation of efficacy of balloon inflation on venous cannulation pain in children: a prospective, randomized, controlled study. Anesth Analg. 2006 May;102(5):1372-5. doi: 10.1213/01.ane.0000205741.82299.d6. PMID 16632812
- [Background] Usichenko TI, Pavlovic D, Foellner S, Wendt M. Reducing venipuncture pain by a cough trick: a randomized crossover volunteer study. Anesth Analg. 2004 Feb;98(2):343-345. doi: 10.1213/01.ANE.0000094983.16741.AF. PMID 14742367
- [Background] Wallace DP, Allen KD, Lacroix AE, Pitner SL. The "cough trick:" a brief strategy to manage pediatric pain from immunization injections. Pediatrics. 2010 Feb;125(2):e367-73. doi: 10.1542/peds.2009-0539. Epub 2010 Jan 11. PMID 20064862